CLINICAL TRIAL: NCT04468256
Title: The Heart Hive COVID-19 Study: A Longitudinal Observational Study of the Impact and Clinical Outcomes of the COVID-19 Pandemic on Individuals With Heart Muscle Disease
Brief Title: The Heart Hive COVID-19 Study
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 20IC6036
Record Dates: First submitted 2020-07-09; First posted 2020-07-13 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: COVID-19; Cardiomyopathies
Keywords: COVID-19; cardiomyopathy; HCM; DCM
MeSH Terms: conditions — COVID-19; Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiomyopathy: Heart Hive registered participants with self-reported cardiomyopathy
  Interventions: Other: COVID-19 experience surveys
- Participants without Heart Disease: Heart Hive registered participants without cardiomyopathy or other heart disease.
  Interventions: Other: COVID-19 experience surveys

INTERVENTIONS:
Other: COVID-19 experience surveys — Serial online surveys recording experiences of the COVID-19 pandemic.

SUMMARY:
All patients with heart disease should have the opportunity to participate in research into their condition, to advance knowledge and treatment.

The HeartHive COVID-19 study is an international online pilot observational cohort study evaluating the impact and clinical outcomes of the COVID-19 pandemic on subjects enrolled in the HeartHive.

Cardiomyopathies are progressive diseases, and there is a need to better understand what factors affect the chances of developing cardiomyopathy, and how the condition progresses.

The impact of the COVID-19 pandemic on patients with cardiomyopathy has not been explored and represents a critical unmet need. Insights into exposure, healthcare outcomes, behavioural changes and the psychosocial ramifications of the pandemic are required to better understand the health needs of this population during these unprecedented circumstances and to adapt clinical services to meet these.

The study will entail completing serial online surveys during the pandemic.

This study uses The Heart Hive - an international, online registry of patients with self-reported clinically diagnosed cardiomyopathy, and people without heart disease. Participants enrol and upload their own data through the website. It is the second research study that will be offered to registry participants and delivered through The Heart Hive platform.

DETAILED DESCRIPTION:
The impact of the COVID-19 pandemic on patients with cardiomyopathy has not been explored and represents a critical unmet need. Insights into exposure, healthcare outcomes, behavioural changes and the psychosocial ramifications of the pandemic are required to better understand the health needs of this population during these unprecedented circumstances and to adapt clinical services to meet these.

The requirements for the population to limit social interaction and stay at home significantly limits conventional research approaches to studying the effect of the pandemic on patients. The Heart Hive platform circumnavigates this by offering an online mechanism to gain insight into the effect of the pandemic in a pre-assembled cohort of patients rapidly and in real-time as the pandemic evolves without any risk to patients.

This study is framed around the following hypotheses:

1. Patients with cardiomyopathy who contract COVID-19 are at greater risk or death or hospitalisation than subjects without heart disease.
2. Patients with cardiomyopathy perceive themselves to be at enhanced risk and are more likely to be following national recommendations on social restriction measures than subjects without heart disease.
3. Patients with cardiomyopathy have experienced interruption to the delivery of their usual cardiology/cardiomyopathy clinical service as a result of the pandemic.
4. Patients with cardiomyopathy are less likely to seek medical help due to fear of contracting COVID-19.
5. The psychological impact of the pandemic is greater in patients with cardiomyopathy than in subjects without heart disease.

Primary Objectives:

1. To conduct serial surveys in patients with cardiomyopathy and subjects without heart disease evaluating the health-related, behavioural and psychosocial impact of the COVID-19 pandemic.
2. To use national registries, including NHS Digital, Office for National Statistics (ONS), Hospital Episodes Statistics (HES) and medical records to longitudinally assess hospital admissions and patient mortality from COVID-19 for UK-based participants.

Secondary Objectives:

1. To use serial surveys to evaluate the indirect impact of COVID-19 on access to healthcare amongst patients with cardiomyopathy.

The Heart Hive COVID-19 study is an international online pilot observational cohort study evaluating the impact and clinical outcomes of the COVID-19 pandemic on subjects enrolled in the Heart Hive. Patients with heart muscle disease and subjects without heart disease who are Heart Hive registry members are eligible to enrol. Eligible subjects who provide informed consent will be enrolled. The study will entail completing serial online surveys during the pandemic. For subjects who live in the UK who provide consent, health information and outcome data will also be collected from NHS digital, national registries (e.g. ONS, HES, DID) and medical records.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and over) Males or Females
* Capacity to provide informed consent
* Subjects with either:

  * A self-reported confirmed diagnosis of cardiomyopathy (dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic cardiomyopathy, restrictive cardiomyopathy, left ventricular non-compaction cardiomyopathy) Or
  * No self-reported history of heart disease

Note: Pregnant women are eligible. This study is observational and entirely separate from clinical care.

Exclusion Criteria:

- Patients who lack capacity to consent for themselves Vulnerable groups (e.g. those under 18, prisoners, those in a dependent relationship, the mentally ill)

- Although usually considered a vulnerable group, pregnant women are eligible for this study which is observational and entirely separate from clinical care.

Patients with a confirmed history of coronary artery disease:

* who have been informed by their treating physician that their cardiomyopathy is secondary to their coronary artery disease, or
* who have undergone previous percutaneous coronary intervention or coronary bypass surgery History of primary valvular heart disease or congenital heart disease Severe, untreated or untreatable hypertension (systolic blood pressures routinely >180 mm Hg and/or diastolic blood pressures >120 mm Hg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart Hive registry members with cardiomyopathy and subjects without heart disease will be invited to enrol in the Heart Hive COVID-19 study. All registry members have previously given consent to be invited by members of the study team to participate in future studies and understand that this is voluntary. The Heart Hive COVID-19 study may be advertised on social media (including Twitter, Facebook and Instagram). The study team may advertise the study via adverts placed with medical society and patient organisation magazines and websites (e.g. Cardiomyopathy UK and Pumping Marvelous).
  There is no limit on the number of participants in the study. This reflects the pilot design of the project and the flexibility afforded by the online platform via which the study is delivered.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2020-07-26 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Qualitative measures of exposure, perception of risk, behaviour, and experience during the COVID-19 pandemic. | 2 years
  Collected from serial online surveys
Health Outcomes | 2 years
  Hospital admissions and deaths due to COVID-19, incidents of major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: James S Ware, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only de-identified data may be shared with other researchers

REFERENCES:
- [Derived] Hammersley DJ, Buchan RJ, Lota AS, Mach L, Jones RE, Halliday BP, Tayal U, Meena D, Dehghan A, Tzoulaki I, Baksi AJ, Pantazis A, Roberts AM, Prasad SK, Ware JS. Direct and indirect effect of the COVID-19 pandemic on patients with cardiomyopathy. Open Heart. 2022 Jan;9(1):e001918. doi: 10.1136/openhrt-2021-001918. PMID 35086919
- See also: The Heart Hive — https://www.thehearthive.org/

DOCUMENTS (1):
  • Informed Consent Form (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT04468256/ICF_000.pdf